CLINICAL TRIAL: NCT03624803
Title: Usage of Dapagliflozin - a Sodium Glucose Co-transporter Inhibitor, in the Management of Type-2 Diabetes Mellitus: A Real World Evidence Study in Egyptian Patients
Brief Title: DAPA - Egypt Study
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1690R00049
Record Dates: First submitted 2018-07-30; First posted 2018-08-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Type-2 Diabetes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Approximately 39 million people of adults aged 20-79 are living with Diabetes in MENA region in 2017, Egypt is number 8 in the top 10 countries in number of adults with Diabetes (8.2 million), where Egypt represents 21% of the Diabetics in MENA region.

Metformin is used as 1st line oral anti-diabetic drug in most cases. Sulfonylureas (SU) are used as frequent first add-on after failure of metformin monotherapy. Sodium Glucose Co-transporter 2 (SGLT2) inhibitors are a newer class of therapy which has a lower incidence of hypoglycemia and in addition helps in weight and BP reduction. In Egypt, SGLT2 inhibitors were introduced in 2016. It is not yet widely used for various reasons including lack of wide clinical experience in Egyptian patients and safety concerns particularly related to infections and some rare Diabetic Ketoacidosis (DKA). Also, usage of SGLT2 inhibitors is limited in the early stage of diabetes as they are usually preferred as 3rd or 4th add-on therapy.

The existing dapagliflozin phase-3 clinical trial program on SGLT2 inhibitors didn't include subjects from Egypt. There is no study available which evaluates the effect of dapagliflozin in real world scenario in Egypt. Key opinion leaders in diabetes in Egypt have also identified the need for study on Egyptian subjects to observe the usage pattern and effect of dapagliflozin, a SGLT2 inhibitor, in this specific real world setting. Therefore, there is a need for data on real world setting across Egypt. With this aim in mind, the present study has been planned.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with 18 years and above.
2. Patients who provide written informed consent.
3. Patients with previously diagnosed Type-2 diabetes mellitus
4. Patients with inadequately controlled diabetes (HbA1c>7%) with existing anti-diabetic medications, prior to initiation of dapagliflozin treatment.
5. Patients who initiated dapagliflozin at least 3 months prior to the date of study start.
6. Patients who are having past medical records for demographic information, weight, blood pressure, HbA1c value, and concomitant medications at the time of dapagliflozin prescribed.

Exclusion Criteria:

1. Patients with Type-1 diabetes mellitus.
2. Patients with any medical condition which in the opinion of the investigator would interfere with safe completion of the study
3. Pregnant or lactating women
4. Patients with other severe conditions/elements which require / may require hospitalization, during study participation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a non-interventional, multi centre, retrospective -prospective, observational study to be conducted at up to 50 sites in Egypt. The study targets to enroll 200 patients. The study would enroll T2DM patients who are/were inadequately controlled (HbA1c >7%) with existing antidiabetic medications and who have been prescribed dapagliflozin at least 3 months prior to study initiation. No study medication will be prescribed or administered as a part of study procedure. Patients, who have been treated as per Investigators' routine clinical practice and prescribed dapagliflozin at least 3 months before will be screened for enrolment in study. Dosage of dapagliflozin and other medications should be as per the routine clinical practice and prescribing information. The study will be initiated after obtaining written approval of Independent Ethics Committee (IEC) /Institutional Review Board (IRB).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-03-09 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
To describe baseline characteristics of patients starting Dapagliflozin together with other anti-diabetic medications , alone or in combination. And to describe if Dapagliflozin was given as 2nd line , 3rd line or later in combination therapy. | 6 months
  To describe baseline characteristics of patients starting Dapagliflozin together with other anti-diabetic medications , alone or in combination. And to describe if Dapagliflozin was given as 2nd line , 3rd line or later in combination therapy.
  "The primary end point will record if Dapagliflozin is used as first or second or third line of treatment.
  also will record if Dapagliflozin used as mono-therapy or in combination with other anti-diabetic medication stating these medications."

SECONDARY OUTCOMES:
To record the mean change in HbA1C from baseline to months 3 and 6. | 6 months
  To record the mean change in HbA1C from baseline to months 3 and 6.
  The Dapagliflozin Egypt's study will enroll patients currently on dapagliflozin at least for 3 months & will follow up these patients for another 3 months, so the total duration is 6 months.
To record the HbA1c change (%) as per different baseline HbA1c levels (<8%, 8-10% and >10%). | 6 months
  To record the HbA1c change (%) as per different baseline HbA1c levels (<8%, 8-10% and >10%).
  "Measurement of HbA1c level (%) change from baseline."
To record percentage of patients achieving HbA1c target (less than or equal 7 %) | 6 months
  To record percentage of patients achieving HbA1c target (less than or equal 7 %).
  "Measurement of percentage of patients achieving HbA1c target less than or equal 7%."
To record the change in weight (kg) as per different baseline BMI (kg/m2) (<25, 25-30, >30). | 6 months
  To record the change in weight (kg) as per different baseline BMI (kg/m2) (<25, 25-30, >30).
  "Measurement the change in weight in Kg from baseline."
To record the change in blood pressure (mmHg) from baseline. | 6 months
  To record the change in blood pressure (mmHg) from baseline.
  "Measurement of blood pressure change from baseline in mmHg."

CONTACTS AND LOCATIONS:
Locations (20):
- Egypt (20):
  - Research Site, Behira, Egypt
  - Research Site, El Rehab, Egypt
  - Research Site, Fiasal, Egypt
  - Research Site, Haram, Egypt
  - Research Site, Madīnat an Naşr, Egypt
  - Research Site, Manial, Egypt
  - Research Site, Mohandesin, Egypt
  - Research Site, Nozha, Egypt
  - Research Site, Sharkia, Egypt
  - Research Site, West Lbalad, Egypt
  - Research Site, Al Mansurah
  - Research Site, Alexandria
  - Research Site, Asyut
  - Research Site, Cairo
  - Research Site, Giza
  - Research Site, Heliopolis
  - Research Site, Maadi
  - Research Site, Mohandessin
  - Research Site, Sohag
  - Research Site, Tanta

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1690R00049&attachmentIdentifier=34556e65-4541-428f-85f8-a73436f45e49&fileName=D1690R00049_CSR_synopsis_redacted.pdf&versionIdentifier=